CLINICAL TRIAL: NCT01214330
Title: A Pilot Study for a Non-Inferiority Trial of Clinician-Collected Versus Patient-Collected Cervical Papanicolaou Smears
Brief Title: Clinician-Collected Versus Patient-Collected Cervical Pap Smears
Acronym: SoloPaP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FWH20100177H
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient-Collected Cervical Pap Smear (Experimental): women will receive a self Papanicolaou Smear test (SoloPap) in addition to their physician-collected Papanicolaou Smear
  Interventions: Device: Patient-Collected Cervical Pap Smear

INTERVENTIONS:
Device: Patient-Collected Cervical Pap Smear — Patient-Collected Cervical Papanicolaou Smear
  Other Names: SoloPap

SUMMARY:
The purpose of this study is to see if it is possible to conduct a full study to determine whether the SoloPap™ cervical cell sample collection kit is as good as a clinician performed Pap test in detecting precancerous cervical lesions in females.

Begin to determine patient attitudes regarding ease of use and discomfort using SoloPap.

DETAILED DESCRIPTION:
The SoloPap "kit" provides to subjects who would not otherwise have a Pap smear done a convenient and private way to collect samples and ship them to a laboratory for processing. The current study is pilot/pre-cursor study for a larger subsequent study that aims to determine whether SoloPap is truly noninferior to clinician-collected Pap smears in detecting cervical pathology. It will also determine user preference and willingness to perform a self- test.

ELIGIBILITY:
Inclusion Criteria:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* All women at least 18 yrs of presenting for Pap Smear who have not previously participated in this protocol. SoloPap can be performed any day that a woman is not having vaginal bleeding

Exclusion Criteria:

* Age <18 years (not recommended for Pap Smear)
* Known pregnancy
* Women who have had a total hysterectomy (cervix removed)
* Women with vaginal bleeding
* Persons who report a history of severe neuropathy or arthritis of the hands or those having other major problems with dexterity of the hands

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, M.D., Principal Investigator — Mke O'Callaghan Federal Hospital
Locations (1):
- Mike O'Callaghan Federal Hospital/Nellis Air Force Base, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 females, age >18, without severe hand arthritis were recruited at the Mike O'Callaghan Military Medical Center (formerly Mike O'Callaghan Federal Hospital). The first participant was enrolled January 19, 2011 and the last patient enrolled was September 1, 2011.
Pre-assignment Details: Of the 150 participants enrolled, 146 participants received all study interventions (comparison of a self-collected Pap smear with Physician-collected samples).
Groups:
- Self Pap Smear and Physician Collected Pap Smear: (solopap) self-collected Pap smear and Physician-collected samples.
Period: Overall Study
Arm/Group | Self Pap Smear and Physician Collected Pap Smear
Started | 150
Completed ((Analyzed)) | 146
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 146 females, age >18
Groups:
- Solopap and Physician-collected Pap Smear: females, age >18, without severe hand arthritis
Arm/Group | Solopap and Physician-collected Pap Smear
Number analyzed (Participants) | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 146
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Pap Test Results Between Self- and Physician-collected Pap Tests
Description: whether the SoloPap™ cervical cell sample collection kit used by the subject (patient) is as good as a clinician performed Pap test in detecting precancerous cervical lesions in females.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Self Pap Smear and Physician Collected Pap Smear
Number analyzed (Participants) | 102
Participants
  positive+positve | 8
  negative+negative | 89
  positive MD + negative solo | 2
  positive solo+negative MD | 3

2. Secondary Outcome: Patient Opinions
Description: Results from a survey about simple subject attitudes regarding the SoloPap.
  Patient Solo Pap Kit Questions
  1. Did you experience any discomfort while using the Solo Pap Kit? Yes / No
  2. Would you use the Solo Pap Kit for future Pap Tests? Yes / No
  3. Would you recommend the Solo Pap Kit to a friend or family member? Yes / No
Time Frame: Directly after interventions (Solo Pap and physician-collected pap smear samples)
Population: 146 females recruited from an outpatient clinic in a military treatment facility, age >18, without severe hand arthritis who completed both the Solo Pap and physician-collected pap smear.
Measure: Count of Participants; unit: Participants
Groups:
- SoloPap Attitude: 1. Did you experience any discomfort while using the SoloPap Kit? (YES/NO)
  2. If you answered yes to the above question how would you describe your discomfort; (MILD/MODERATE/SEVERE)
  3. Would you use the SoloPap Kit for future Pap Tests? (YES/NO)
  4. Would you recommend the SoloPap Kit to a friend or family member? (YES/NO)
Arm/Group | SoloPap Attitude
Number analyzed (Participants) | 146
Participants
  discomfort while using solopap: yes | 36
  discomfort while using solopap: no | 65
  discomfort while using solopap: no response | 45
  use solopap in future: yes | 91
  use solopap in future: no | 11
  use solopap in future: no response | 44
  recommend solopap: yes | 97
  recommend solopap: no | 4
  recommend solopap: no response | 45

ADVERSE EVENTS:
Time Frame: 1 hour for each participant during pap procedures.
Groups:
- Self Pap Smear: SoloPap: Patient-Collected Cervical Papanicolaou Smears
  Self Pap Smear
Arm/Group | Self Pap Smear
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

LIMITATIONS AND CAVEATS:
Limitations:

Higher socioeconomic status of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2011-08-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT01214330/ICF_000.pdf